CLINICAL TRIAL: NCT06516016
Title: Multimodal Markers of Neurodegenerative Disorders at Presymptomatic Stages
Acronym: NEUROPREMS
Status: Not yet recruiting | Type: Observational
Sponsor: Paris Brain Institute (ICM) (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A00824-43
Record Dates: First submitted 2024-06-06; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases | interventions — Posture; Blood Specimen Collection; Spinal Puncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 800 presymptomatic participants: * Visit interview
  * Neurological evaluation (NeuroPrems Scale and Self-administered REDCap questionnaires)
  * Psychological evaluation (Motivation, life trajectories and experiencies and semi-structured interview)
  * Cognition and behavior evaluation (Neuropsychological battery and Self-administered REDCap QR)
  * Imaging (MRI 3T and PET DPA-714)
  * Neurophysiology (Eye movement recording, Magnetoencephalography, Body posture and gait recording, voice and language recording)
  * Skin aging (Skin quantitative elasticity assessment)
  * Sleep (Videopolysomnography)
  * Biosampling (Blood draw, lumbar puncture, saliva sampling, skin biopsy, nasal brush and tear fluid collection)
  Interventions: Radiation: PET; Other: MRI 3T; Other: Oculomotricity assessment; Other: Magnetoencephalography assessment; Other: Body posture and gait assessment; Other: Voice recording; Other: Video-polysomnography; Biological: Blood sampling, skin biopsy, excreta sampling, lumbar puncture
- 200 healthy volunteers: * Visit interview
  * Neurological evaluation (NeuroPrems Scale and Self-administered REDCap questionnaires)
  * Psychological evaluation (Motivation, life trajectories and experiencies and semi-structured interview)
  * Cognition and behavior evaluation (Neuropsychological battery and Self-administered REDCap QR)
  * Imaging (MRI 3T and PET DPA-714)
  * Neurophysiology (Eye movement recording, Magnetoencephalography, Body posture and gait recording, voice and language recording)
  * Skin aging (Skin quantitative elasticity assessment)
  * Sleep (Videopolysomnography)
  * Biosampling (Blood draw, lumbar puncture, saliva sampling, skin biopsy, nasal brush and tear fluid collection)
  Interventions: Radiation: PET; Other: MRI 3T; Other: Oculomotricity assessment; Other: Magnetoencephalography assessment; Other: Body posture and gait assessment; Other: Voice recording; Other: Video-polysomnography; Biological: Blood sampling, skin biopsy, excreta sampling, lumbar puncture

INTERVENTIONS:
Radiation: PET — [18F]DPA-714 will be injected intravenously as a 1 minute intravenous bolus injection and dynamic PET acquisition will last 90 min. The aim is the quantification of the neuroimmune reaction during neuroinflammation process.
Other: MRI 3T — Brain MRI will aim at providing imaging biomarkers which will allow evaluating brain structure, microstructure, iron load, myelin, neurodegeneration of the substantia nigra and locus coeruleus, functional connectivity, brain perfusion and the glymphatic system.
Other: Oculomotricity assessment — Recording eye movements in a controlled environment (requiring no specific room or area) in binocular vision at a frequency > 500Hz, while retaining infrared video footage of eye movements for high-quality clinical monitoring.
Other: Magnetoencephalography assessment — Recording brain magnetic activity using the Elekta Neuromag® TRIUX Magnetoencephalograph ; The participant will be comfortably seated in an adjustable-height chair. The device is enclosed in a shielded room isolated from external electric and magnetic fields to measure the extremely weak magnetic activities produced by the brain.
Other: Body posture and gait assessment — The acquisition of kinematic gait parameters will be achieved ; markers are positioned on the different segments of members, recognized by a camera system positioned on the walls. Neurophysiologic muscular activity of the lower limbs will also be recorded.
Other: Voice recording — Participants will be recorded during a single session at every visit upon baseline with a professional quality head mounted microphone.
Other: Video-polysomnography — Participants will complete standard sleep questionnaires before the visit and perform neurophysiological tests including cognitive tasks before and after the sleep recording.
Biological: Blood sampling, skin biopsy, excreta sampling, lumbar puncture — Experimental analyses, genetic and multi-OMIC analyses for biomarker research.

SUMMARY:
NeuroPrems is a prospective, monocentric, longitudinal, not relating to a medicinal product for human use, non-randomized, non-controlled research. The study mainly aims to identify longitudinal changes and events in multimodal markers of neurodegeneration and neuroinflammation during the presymptomatic phases of neurodegenerative diseases.

ELIGIBILITY:
1. Inclusion Criteria :

   1. For all participants :

      * Male or female
      * Age ≥ 18 years
      * Signed Informed consent by the subject
      * Affiliated with a social security system or beneficiary of such a regime
      * Ability to undergo an MRI exam with Gadobutrol
   2. For presymptomatic participants only :

      * Absence of a diagnosis of neurodegenerative disease. And at least one of the criteria :
      * Known carrier or relative of a patient carrying a mutation in a causal or at-risk responsible for a neurodegenerative disease
      * Isolated REM sleep behavioral disorder
      * Radiological isolated syndrome
      * Abnormal brain protein aggregates
   3. For controls only :

      * Absence of symptoms or diagnosis of neurodegenerative disease (or criteria corresponding to at risk group)
2. Exclusion Criteria :

   * Clinical symptoms fulfilling the criteria of a neurodegenerative disease (see table in criteria section)
   * Refusal of blood draw or brain MRI
   * MRI contraindication (see criteria section)
   * Known allergy to gadoteric acid
   * Unwillingness to be informed in case of abnormal MRI (with a significant medical anomaly)
   * Pregnancy or breastfeeding. For women in fertile age a urine pregnancy test will be performed before the MRI.
   * Inability to understand information about the protocol
   * Person deprived of their liberty by judicial or administrative decision
   * Person under legal protection (legal guardianship, tutelage or maintenance of justice)
   * Person without any protection and unable to consent
   * Other medical, neurological, psychiatric, or social conditions that in the investigator's opinion are likely to interfere with study conduct.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will focus on subjects potentially at high risk of developing a degenerative disease, compared to a control population of healthy volunteers and relatives with no evidence of genetic mutation under study, radiologically isolated syndrome (RIS), Idiopathic rapid eye-movement (REM) sleep behavior disorder (iRBD) and abnormal elevated levels of protein ptau217.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2034-08-31 (Estimated); Study Completion 2034-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of change of clinical, neurophysiological, anatomical and molecular marker profiles of neurodegenerescence and neuroinflammation in presymptomatic individuals | Baseline, Year 1, Year 2, Year 3, Year 4 and Year 5
  Clinical markers will be: neurological and neuropsychological testing, and questionnaires; Neurophysiological markers will link functional brain networks and cognitive processes by using MEG, kinematic or eye movement recordings; Anatomical markers will be: cerebral MRI, glymphatic imaging, PET and skin elasticity; Molecular markers will be: blood, CSF, skin cells, iPSC derived biomarkers, transcriptomic, proteomic and metabolomic signatures

SECONDARY OUTCOMES:
Intra-individual change in trajectory profiles determined by multimodal analysis | Baseline, Year 1, Year 2, Year 3, Year 4 and Year 5
  Determination by individual parameters form multimodal analysis
Rate and mean time to symptomatic conversion/progression | Baseline, Year 1, Year 2, Year 3, Year 4 and Year 5
  Conversion/progression defined according to international criteria for the clinical diagnosis of each disease
Mean time of onset in genetically presymptomatic individuals | Baseline, Year 1, Year 2, Year 3, Year 4 and Year 5
  Estimated time to onset in genetic presymptomatic individuals from the average age at diagnosis among affected family members
Rate of change for each study marker | Baseline, Year 1, Year 2, Year 3, Year 4 and Year 5
  Period of changes defined (1) as breakpoints in the longitudinal evolution; (2) early, intermediate or late progression for each marker in the whole cohort and for each pathological group
Rate of change in the self-administered questionnaires | Baseline, Year 1, Year 2, Year 3, Year 4 and Year 5
  Changes in the self-administered questionnaires on motivation, barriers and psychology
Rate of change in consumption of information issued from Consultations, hospitalizations and medication prescriptions | From Year -10 to Year 10 (annual update)
  Data from SNDS will be extracted during a 10-year period before and 10-year after the cohort entry. This follow-up should allow for a better understanding of when conversion occurs and to compare pathologies which involve a fairly broad spectrum of evolution.
Time to loss of autonomy | Baseline, Year 1, Year 2, Year 3, Year 4 and Year 5
  Rate of change from baseline of at least 0.1 in the utility index from EQ-5D-51

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No